CLINICAL TRIAL: NCT01269151
Title: A Prospective, Non-randomized, Mono-center, Cohort Study to Evaluate the Short- and Long-term Effects of 0.5mg Intraocular Ranibizumab (Lucentis) Injections on Retinal Function in Patients With Wet Age-related Macular Degeneration During Twelve Month
Brief Title: Ranibizumab Short- and Log-term Effects on Retinal Function in wAMD
Acronym: LucERG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Dr. Matthias Lueke, Dr. med. Matthias Lüke, University of Luebeck
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LucERG-001
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Age-Related Macular Degeneration; Retinal Function
Keywords: Age-Related Macular Degeneration; Retinal Function; multifocal-ERG; Electroretinography; microperimetry; Lucentis; Ranibizumab; longterm effects; best corrected visual acuity; BCVA
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lucentis (Ranibizumab) (Experimental)
  Interventions: Drug: Lucentis (Ranibizumab)

INTERVENTIONS:
Drug: Lucentis (Ranibizumab) — Ranibizumab Short- and Log-term Effects on Retinal Function measured by Multifocal-ERG and Microperimetry

SUMMARY:
Multifocal-electroretinoram (ERG) and microperimetry are objective criteria to asses retinal function. No information besides visual acuity exist for the development of retinal function during the course of wet AMD during therapy with Lucentis. The aim of our study is to evaluate the value of multifocal-ERG and microperimetry as an sensitive tool and early predictor of recurrence of the disease. The second goal will be to evaluate the neuroprotective effects of an adequate therapy on retinal function using microperimetry and multifocal-ERG during the course of wet AMD.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients above 50 years of age
2. wet age-related macular degeneration (AMD)
3. an available follow-up of 12 months
4. written informed consent
5. visual acuity of 0.1 or better

Exclusion Criteria:

Systemic conditions or treatments

1. history or evidence of severe cardiac disease (e.g., NYHA functional class III or IV)
2. clinical or medical history of unstable angina, acute coronary syndrome, myocardial infarction or revascularization within the last 6 months
3. ventricular tachyarrythmias requiring ongoing treatment
4. History or evidence clinically significant peripheral vascular disease, such as intermittent claudication or prior amputation
5. Clinically significant impaired renal or hepatic function
6. Stroke within 12 month before trial entry.
7. Known serious allergies to the fluorescein dye use in angiography
8. Known contraindications to the components of Lucentis® formulation.

Ocular concomitant conditions/ diseases

1. Active intraocular inflammation (grade trace or above) in either eye
2. Any active infection (e.g. conjunctivitis, keratitis, scleritis, uveitis, endophthalmitis) in either eye
3. History of uveitis in either eye
4. Treatment with anti-angiogenic drugs (pegaptanib sodium, anecortave acetate,bevacizumab, etc.) or intravitreal corticosteroids in either eye within 3 months prior to inclusion
5. Angle block glaucoma
6. Phthisis
7. Intraocular Pressure <10mmHg
8. Macular or retinal dystrophies

Compliance/ Administrative

1. Previous participation in any clinical studies of investigational drugs (excluding vitamins and minerals) within 1 month (or a period corresponding to 5 half-lives of the investigational drug, whatever is longer) prior to inclusion.
2. Patients will be excluded who were younger than 50 years according of the definition of age-related AMD.
3. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant.
4. Pregnant or nursing (lactating) women
5. Inability to comply with study or follow-up procedures.
6. Any treatment with an investigational agent in the past 3 months any condition.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2013-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Changes of retinal function of the macula monitored by multifocal-ERG and microperimetry as measured 12 months. | 12 months
  Main outcome measures are the changes of retinal function of the macula monitored by multifocal-ERG and microperimetry as measured 12 months.

SECONDARY OUTCOMES:
to document changes in best corrected visual acuity (BCVA) measured on 4 meters, | 12 months
  to document changes in best corrected visual acuity (BCVA) measured on 4 meters,
to document changes in angiography | 12 months
  to document changes in angiography
to document changes in optical coherence tomography (OCT) | 12 months
  to document changes in optical coherence tomography (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Grisanti, M.D. Prof., Principal Investigator — University of Luebeck - Department of Ophthalmology: Germany
Locations (1):
- University of Luebeck - Department of Ophthalmology, Lübeck, Germany

REFERENCES:
- See also: University of Luebeck - Department of Ophthalmology - Germany — http://www.uksh.de/Augenklinik_Luebeck/index.html